CLINICAL TRIAL: NCT05931471
Title: Effect of Yogurt on Mucosal Immunity in the Gastrointestinal Tract
Brief Title: Yogurt and GI Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FL119
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Yogurt Intake; Gastrointestinal Immune Function; Gut Microbiome; Gut Health
Keywords: Yogurt; Adults; Gut microbiome; Gut health; Immune function; GI tract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yogurt Consumption (Experimental): Participants will complete a 2-week baseline with no yogurt intake, followed by a three-week yogurt intervention, and then a 2-week follow-up period with no yogurt intake.
  Interventions: Other: Yogurt Intervention

INTERVENTIONS:
Other: Yogurt Intervention — Participants will be provided with a commercial yogurt that contains only cultured dairy, traditional live active cultures (Streptococcus thermophilus, Lactobacillus delbrueckii subsp. bulgaricus, and possibly other non-brand-specific strains), sugar, and, optionally, vanilla flavor. The yogurt will contain no starches or pectin, gums, fiber or other added ingredients. Participants will be asked to consume two 6-ounce portions of yogurt each day, and to log their consumption in a provided booklet. They will be advised to incorporate the yogurt into their diet however they choose (as part of meals or as snacks), to avoid other fermented foods, and to otherwise maintain their habitual diet.

SUMMARY:
The purpose of this research is to assess mucosal immune function responses in the gastrointestinal (GI) tract to twice-daily yogurt consumption. Previous research has shown that dairy yogurt intake can benefit gastrointestinal health. The current study will determine whether a dietary intervention with dairy yogurt will improve mucosal immunity and the gut microbiome.

DETAILED DESCRIPTION:
The gastrointestinal (GI) tract has the difficult task of absorbing nutrients while excluding microorganisms and non-nutritive foreign agents. The GI tract is protected by components of GI mucosal immunity, such as the mucin layer, anti-microbial peptides, secretory IgA (sIgA), and more, which collectively maintain gut homeostasis. When mucosal immunity fails, the result can be gastrointestinal infection, allergic inflammation, or inflammatory bowel disease. Mechanistic knowledge from in vitro studies suggests that sIgA increases in response to lactic acid bacteria and mucin-2 expression increases in response to milk peptides in yogurt. Yogurt consumption may also reduce constipation and increase the production of short-chain fatty acids (SCFAs). SCFAs promote the health of intestinal cells by acting as an energy source, influencing gene expression, and exerting anti-inflammatory effects. When SCFAs increase, fecal pH decreases.

This research will expand the limited existing literature on how GI mucosal immunity changes in response to yogurt consumption, the time frame over which effects occur and how long the effects persist after yogurt is discontinued. Participants will undergo a two-week baseline period without yogurt intake, followed by a three-week intervention of two daily 6-oz servings of dairy yogurt, and a follow-up period with no yogurt consumption. Stool samples will be collected at the end of the 2-week baseline period, after 1, 2, and 3 weeks of intervention, and at the end of the 2 weeks post-intervention period for measurement of fecal sIgA, fecal mucin-2 mRNA, fecal pH, and fecal SCFAs, and analysis of the fecal microbiome. 24-hour dietary recalls will be collected with the Automated Self-Administered Dietary Assessment Tool (ASA24) during the baseline and intervention phases of the trial.

Specific knowledge will be produced regarding the effect of regular yogurt consumption on sIgA levels, mucin-2 gene expression and fecal pH in older adults (age 50 - 75 years). The study will also produce knowledge on the intervention length needed for maximal response in these outcome measures and how long these responses persist when the yogurt intervention is discontinued. The outcomes of this study will 1) provide preliminary data to inform design of future, larger studies on how dairy yogurt or similar cultured products influence GI mucosal immune function, and 2) contribute to growing knowledge on the potential health benefits of consuming fermented, particularly yogurt.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 - 75 years
* BMI 18.5 - 39.9 kg/m2

Exclusion Criteria:

* BMI less than 18.5 or greater than 39.9
* Consumption of fermented foods or probiotics in the past two weeks
* Unwillingness to abstain from non-study fermented foods and probiotics during the trial
* Allergy to cow milk
* Lactose intolerance
* Any dietary restriction limiting or prohibiting consumption of lightly sweetened, vanilla flavored, whole milk yogurt
* Uncomfortable with or unwilling to complete stool sample collections
* Current participation in another research study
* If female,

  * Currently pregnant or lactating
  * Have had menstrual bleeding in the past 12 months
* Having fewer than 3 bowel movements per week
* Unmanaged hypertension, defined as blood pressure greater than or equal to 140/90 mmHg
* Current diagnosis of:

  * Disease that affects the immune system, including HIV/AIDS
  * Cancer
  * Diabetes
  * Asthma with daily medication
  * Primary immune deficiency
  * Auto-immune disease
  * Chronic gastrointestinal disorder (e.g. Crohn's disease, irritable bowel syndrome, colitis, gastric ulcer)
* Current use for 2 weeks or longer of:

  * Any drug that affects the immune system, such as immunosuppressants, immune modifying drugs, or corticosteroids (e.g. cortisone, prednisone, methylprednisolone)
  * Biologics (e.g. Lantus, Remicade, Rituxan, Humira, Herceptin, Avastin, Lucentis, Enbrel)
* Use of sulfonamides or antibiotics in the past 3 months
* Use of laxatives in the past 2 weeks
* Currently undergoing cancer treatment with radiation or drugs
* History of gastrointestinal surgery that would impact study outcomes, such as gastric bypass, intestinal resection, surgeries of the liver or pancreas, or removal of part or all of any organ of the GI tract
* Having within the past 2 weeks:

  * Diarrheal illness, defined as passing 3 or more abnormally loose or watery stools in a 24-hour period
  * Persistent vomiting
  * Fever
* Having within the past 3 months:

  * Surgery
  * Hospitalization
* Having within the past 1 month:

  * Colonoscopy

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Changes in fecal secretory immunoglobulin A | At end of 2-week baseline period; at 1, 2 and 3 weeks of intervention; and at end of 2-week follow-up period
  Fecal secretory immunoglobulin A (sIgA) will be extracted then measured in duplicate by enzyme-linked immunosorbent assay (ELISA)

SECONDARY OUTCOMES:
Changes in fecal mucin-2 mRNA expression | At end of 2-week baseline period; at 1, 2 and 3 weeks of intervention; and at end of 2-week follow-up period
  Pre-amplification and quantitative reverse transcription polymerase chair reaction (RT-qPCR) for mucin 2 (MUC2) and GAPDH will be conducted using validated TaqMan assays, and fold MUC2 gene expression of samples will be calculated relative to a commercial total human colon RNA standard using GAPDH as the housekeeping gene.
Changes in fecal pH | At end of 2-week baseline period; at 1, 2 and 3 weeks of intervention; and at end of 2-week follow-up period
  Fecal pH will be measured with a glass electrode pH meter.
Changes in fecal short-chain fatty acids | At end of 2-week baseline period; at 1, 2 and 3 weeks of intervention; and at end of 2-week follow-up period
  The most abundant fecal SCFAs, such as acetate, propionate, butyrate, will be analyzed via gas chromatography-mass spectrometry.
Fecal microbiome | At end of 2-week baseline period; at 1, 2 and 3 weeks of intervention; and at end of 2-week follow-up period
  Gut microbiota composition will be assessed with PCR amplification and 16S sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Danielle G Lemay, PhD, Principal Investigator — USDA, Western Human Nutrition Research Center; Bess L Caswell, PhD, Principal Investigator — USDA, Western Human Nutrition Research Center
Locations (1):
- USDA Western Human Nutrition Research Center, Davis, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared at the time of study publication in accordance with US Department of Agriculture (USDA) policy.
Time Frame: At the time of study publication, de-identified IPD will be permanently archived on a publicly accessible platform.
Access Criteria: De-identified IPD and supporting information will be publicly available.

DOCUMENTS (1):
  • Informed Consent Form (2023-08-04): https://cdn.clinicaltrials.gov/large-docs/71/NCT05931471/ICF_001.pdf